CLINICAL TRIAL: NCT06608563
Title: The Effect of an Adhesive System on the Retention and Caries Prevention for Fissure Sealants in Permanent Molars: a 2-year Randomised Clinical Trial
Brief Title: The Effect of an Adhesive System on the Retention and Caries Prevention for Fissure Sealants in Permanent Molars
Acronym: ResinFS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, Rona Leith, Assistant Professor, University of Dublin, Trinity College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 231104_ResinFS
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Dental Caries; Fissure Sealant
Keywords: fissure sealant; first permanent molar; retention; adhesive system; children; clinical trial; caries
MeSH Terms: conditions — Dental Caries | interventions — Pit and Fissure Sealants

STUDY DESIGN:
Intervention Model Description: Double-blind 2-arm parallel controlled randomised clinical trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcome assessor (independent examiner) and participants will be blind to study groups.
  It is not possible to blind the operator due to differences in material capsule colours/consistency at the time of fissure sealant placement.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fissure sealant without adhesive system (NO BOND) (Active Comparator): Teeth randomised to the control group will be using issure sealant without adhesive system (NO BOND)
  Interventions: Procedure: Fissure sealant without adhesive system (NO BOND)
- Fissure sealant with adhesive system (BOND) (Experimental): Teeth randomised to the test group will be treated using fissure sealant with adhesive system (BOND)
  Interventions: Procedure: Fissure sealant with adhesive system (BOND)

INTERVENTIONS:
Procedure: Fissure sealant without adhesive system (NO BOND) — 1. Cotton roll isolation
  2. Etching of the enamel surface: 17% phosphoric 15 seconds over the surface to be sealed (Phosphoric etchant gel - Vococid, VOCO)
  3. Washing/drying: a 3-1 syringe will be used to rinse all etch material from the toothsurface.
  4. Sealant application: a light-curing nano-hybrid fissure sealant material (Grandio Seal; VOCO) will be applied using the applicator tip.
  5. Lightcuring: The material will be lightcured for 20 seconds.
  Arms: Fissure sealant without adhesive system (NO BOND)
Procedure: Fissure sealant with adhesive system (BOND) — 1. Cotton roll isolation
  2. Etching of the enamel surface: 17% phosphoric 15 seconds over the surface to be sealed (Phosphoric etchant gel - Vococid, VOCO)
  3. Washing/drying: a 3-1 syringe will be used to rinse all etch material from the toothsurface.
  4. Adhesive system application: the adhesive system (Futurabond, VOCO) single dose capsule will be applied over the surface to be sealed for 5 seconds using a microbrush. The adhesive system will be air thin dried and lightcured for 10s before sealant placement.
  5. Sealant application: a light-curing nano-hybrid fissure sealant material (Grandio Seal; VOCO) will be applied using the applicator tip.
  6. Lightcuring: The material will be lightcured for 20 seconds.
  Arms: Fissure sealant with adhesive system (BOND)

SUMMARY:
Background: Resin-based fissure sealants (FS) are recommended to prevent pit-and-fissure caries development or prevent the progression of enamel caries lesion to frank cavitation into dentine. There is still limited clinical evidence on the use of adhesive system beneath fissure sealants in permanent molars and its effect on FS retention and caries progression.

Aim: The aim of this randomised clinical trial is to evaluate the clinical efficacy of fissure sealants placed with and without prior use of an adhesive system in terms of retention and caries prevention in permanent molars over the period of 2 years.

Study design: Children (6-12 years of age) with high caries risk that require sealants in their first permanent molars (ICDAS 0-3) will be selected at the Dublin Dental University Hospital (DDUH). Molars will be stratified according to presence of caries lesions (ICDAS 0 or ICDAS1-3) and randomly allocated according to the study groups (Test group: 17% phosphoric acid + adhesive system + FS; Control group: 17% phosphoric acid + FS). The randomisation unit will be the tooth and more than one tooth can be included per child. All children will be evaluated after 12 and 24 months by calibrated independent examiners. The primary outcome of the present trial is sealant retention over time. Clinical variables such as age, gender, tooth position (upper/lower), caries experience (DMFT/dmft), stage of eruption (erupted/partially erupted) and children's behavior (Frankl scale) will be collected.

DETAILED DESCRIPTION:
Introduction

Resin-based fissure sealants (FS) have been used as a physical barrier in pit-and-fissures with the aim to reduce biofilm accumulation and prevent the development of new caries lesions in first permanent molars. Several international guidelines recommend the use of FS for caries prevention in the paediatric population.

The majority of the FS manufactures recommend the etching of the enamel surface prior to FS application in order to remove any remaining plaque debris and to increase the surface contact area by superficial demineralisation of tooth surface. Resin based-fissure sealants contain light-activated urethane dimethacrylate (UDMA) or bisphenol A-glycidyl methacrylate (Bis-GMA) resin in its composition which bonds to the etched enamel. Several clinical studies have investigated the use of an intermediate layer of adhesive system (primer and bond) in order to increase the bonding strength and increase retention of FS over time in caries free molars, however little is known on the effect on caries progression and the choice of FS protocol for treatment of enamel caries lesions.

Another factor that can influence the performance of resin-based fissure sealant due to hydrophobic characteristics of the material is the presence of saliva contamination (poor moisture control) during application. Therefore, the stage of eruption, patient's behaviour and operator experience can play a major role when it comes to FS retention on tooth surfaces. The majority of clinical trials in the field had trained and experienced operators, including specialists in paediatric dentistry, which could impact the translational and external validity of their findings. More studies are needed with less experienced operators in order to evaluate the effectiveness of FS placement in different environments.

Therefore, the aim of the present randomised clinical trial is to evaluate the effectiveness of resin-based fissure sealant placed by undergraduate dental students with or without an intermediate layer of adhesive system in terms of dentine caries prevention and retention over time.

Methods

Study Design The present study is a two-parallel arm, controlled, single-blind clinical trial. This study will be registered at Clinical Trials website and submitted to approval by the local Ethics Committee (SJH/AMNCH Joint Research Ethics Committee).

Sample Size Calculation For the sample size calculation, we have considered the results of a previous study from McCafferty & O'Connell 2016 (difference of sealant retention between the groups of 13%; bonded 92% and non-bonded 79%). The sample size calculation was performed using https://www.sealedenvelope.com/ website using a significance level of 5% (alpha) and a power of 80% (1-beta). A minimum sample of 112 teeth per group was required. We increased the sample size by 40% to compensate the cluster effect (more than one tooth can be included per child) and possible loss to follow-up. The final sample required is 313 teeth.

Randomisation process The randomisation unit is the tooth and more than one tooth can be included per child. The website https://www.sealedenvelope.com/simple-randomiser/v1/lists will be used for randomisation list generation, using blocks of different sizes (4, 6 and 8). Sealed, sequentially numbered, opaque envelopes will be used and opened at the time of sealant placement.

Operators All sealants will be placed by undergraduate dental students during the undergraduate clinic in Paediatric Dentistry. The treatment will be supervised by an experienced dentist/clinical supervisor.

Interventions

Control group (FS)

1. Cotton roll isolation: cotton roll will be placed buccally and lingually/palatally to the first permanent molar to be treated. A saliva ejector will be used to remove any excess of saliva. If the cotton roll are saturared in saliva at any point of the treatment, they will need to be changed.
2. Etching of the enamel surface: 17% phosphoric acid will be applied for 15 seconds over the surface to be sealed (Phosphoric etchant gel - Vococid, VOCO) using the etch syringe applicator tip.
3. Washing/drying: a 3-1 syringe will be used to rinse all etch material from the toothsurface. A high volume suction will be used. Cotton pellets will be changed to a dry ones at this stage and the surface will be dried for 5s using the air syringe.
4. Sealant application: a light-curing nano-hybrid fissure sealant material (Grandio Seal; VOCO) will be applied using the applicator tip. A probe will be used to ensure that the material is present in all fissures without any air bubbles.
5. Lightcuring: The material will be lightcured for 20 seconds. The material colour will change to an opaque off white colour when exposed to light.
6. Check occlusion: After checking for premature contact points, if there is a need to remove a excess of material, a superfine diamond bur or a silicone finishing point can be used for adjustments.

Test group (Adhesive + FS)

1. Cotton roll isolation: cotton roll will be placed buccally and lingually/palatally to the first permanent molar to be treated. A saliva ejector will be used to remove any excess of saliva. If the cotton roll are saturared in saliva at any point of the treatment, they will need to be changed.
2. Etching of the enamel surface: 17% phosphoric acid will be applied for 15 seconds over the surface to be sealed (Phosphoric etchant gel - Vococid, VOCO) using the etch syringe applicator tip.
3. Washing/drying: a 3-1 syringe will be used to rinse all etch material from the toothsurface. A high volume suction will be used. Cotton pellets will be changed to a dry ones at this stage and the surface will be dried for 5s using the air syringe.
4. Adhesive system application: the adhesive system (Futurabond, VOCO) single dose capsule will be applied over the surface to be sealed for 5 seconds using a microbrush (ative movements along the fissures to ensure bond penetration). The bond will be air thin dried for removal of solvent and excess material. The bond will be lightcured for 10s before sealant placement.
5. Sealant application: a light-curing nano-hybrid fissure sealant material (Grandio Seal; VOCO) will be applied using the applicator tip. A probe will be used to ensure that the material is present in all fissures without any air bubbles.
6. Lightcuring: The material will be lightcured for 20 seconds. The material colour will change to an opaque off white colour when exposed to light.
7. Check occlusion: After checking for premature contact points, if there is a need to remove a excess of material, a superfine diamond bur or a silicone finishing point can be used for adjustments.

Clinical variables such as children's age and gender, tooth position (upper/lower), caries experience (DMFT/dmft), ICDAS score tooth surface (1/2/3), and children's behavior during the procedure (Frankl scale) will be collected.

Evaluations

All children will be evaluated after 12 and 24 months by independent calibrated and blind examiners for both primary (sealant retention) and secondary outcomes.

The presence of dental caries lesion will evaluated according to ICDAS criteria and caries progression into dentine will be recorded. Sealant retention will be evaluated according to the scoring system proposed by Oba et al. 2009: 0 (fully retained sealant); 1 (partially retained sealant) or 2 (absent sealant).

ELIGIBILITY:
Inclusion criteria:

1. 6 to 12 years of age;
2. Referred for dental treatment at the Dublin Dental University Hospital DDUH) or that are ongoing patients of the Paediatric dentistry clinic;
3. With first permanent molars that are caries free or present caries lesions restricted to enamel (ICDAS 1 to 3) indicated for glass ionomer sealants.
4. Whose parents agreed and consent to participate in the present research;

Exclusion criteria:

1. Presence of any developmental defects
2. Presence of any type of restorative/sealant material in the selected tooth;
3. Presence of a dentine shadow (ICDAS 4) or dentine cavitation (ICDAS 5/6) detected clinically and/or radiographically14;
4. Insufficient cooperation to achieve adequate moisture control using cotton roll isolation

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2025-06-05 (Estimated); Study Completion 2027-06-05 (Estimated)

PRIMARY OUTCOMES:
Sealant Retention | Sealant retention will be evaluated after 1 and 2 years.
  Sealant retention will be examined after 1 and 2 years by a trained, calibrated, independent examiner. Sealant retention (secondary outcome) will be evaluated according to the scoring system proposed by Oba et al. 2009: 0 (fully retained sealant); 1 (partially retained sealant) or 2 (absent sealant).
  Early failures will be identified and recorded in the patient's review appointment in the undergraduate clinic.

SECONDARY OUTCOMES:
Caries Progression | Caries Progression will be evaluated after 1 and 2 years
  Caries progression will be examined after 1 and 2 years by a trained, calibrated, independent examiner according to ICDAS criteria (Ismail et al., 2006). Presence of caries progression will be scored if progression into dentine is seen (ICDAS 4-6).
Patient behaviour | Immediately after the procedure
  Patient's behaviour during the treatment will be reported by the operator at the end of the procedure using Frankl's behavior rating scale.

CONTACTS AND LOCATIONS:
Overall Officials: Rona Leith, Principal Investigator — DDUH - Trinity College Dublin
Locations (1):
- Dublin Dental University Hospital - Trintiy College Dublin, Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Memarpour M, Shafiei F, Zarean M, Razmjoei F. Sealing effectiveness of fissure sealant bonded with universal adhesive systems on saliva-contaminated and noncontaminated enamel. J Clin Exp Dent. 2018 Jan 1;10(1):e1-e6. doi: 10.4317/jced.54471. eCollection 2018 Jan. PMID 29670708
- [Background] Nazar H, Mascarenhas AK, Al-Mutwa S, Ariga J, Soparker P. Effectiveness of fissure sealant retention and caries prevention with and without primer and bond. Med Princ Pract. 2013;22(1):12-7. doi: 10.1159/000341155. Epub 2012 Aug 9. PMID 22889920
- [Background] McCafferty J, O'Connell AC. A randomised clinical trial on the use of intermediate bonding on the retention of fissure sealants in children. Int J Paediatr Dent. 2016 Mar;26(2):110-5. doi: 10.1111/ipd.12165. Epub 2015 Apr 10. PMID 25864681
- [Background] Wright JT, Crall JJ, Fontana M, Gillette EJ, Novy BB, Dhar V, Donly K, Hewlett ER, Quinonez RB, Chaffin J, Crespin M, Iafolla T, Siegal MD, Tampi MP, Graham L, Estrich C, Carrasco-Labra A. Evidence-based clinical practice guideline for the use of pit-and-fissure sealants: A report of the American Dental Association and the American Academy of Pediatric Dentistry. J Am Dent Assoc. 2016 Aug;147(8):672-682.e12. doi: 10.1016/j.adaj.2016.06.001. PMID 27470525
- [Background] San Martin-Galindo L, Rodriguez-Lozano FJ, Abalos-Labruzzi C, Niederman R. European Fissure Sealant Guidelines: assessment using AGREE II. Int J Dent Hyg. 2017 Feb;15(1):37-45. doi: 10.1111/idh.12174. Epub 2015 Sep 11. PMID 26359655
- [Background] Welbury R, Raadal M, Lygidakis NA; European Academy of Paediatric Dentistry. EAPD guidelines for the use of pit and fissure sealants. Eur J Paediatr Dent. 2004 Sep;5(3):179-84. No abstract available. PMID 15471528
- [Background] Innes NP, Frencken JE, Bjorndal L, Maltz M, Manton DJ, Ricketts D, Van Landuyt K, Banerjee A, Campus G, Domejean S, Fontana M, Leal S, Lo E, Machiulskiene V, Schulte A, Splieth C, Zandona A, Schwendicke F. Managing Carious Lesions: Consensus Recommendations on Terminology. Adv Dent Res. 2016 May;28(2):49-57. doi: 10.1177/0022034516639276. PMID 27099357
- [Background] van Loveren C, van Palenstein Helderman W. EAPD interim seminar and workshop in Brussels May 9 2015 : Non-invasive caries treatment. Eur Arch Paediatr Dent. 2016 Feb;17(1):33-44. doi: 10.1007/s40368-015-0219-3. Epub 2016 Feb 10. PMID 26860292
- [Background] Schwendicke F, Splieth C, Breschi L, Banerjee A, Fontana M, Paris S, Burrow MF, Crombie F, Page LF, Gaton-Hernandez P, Giacaman R, Gugnani N, Hickel R, Jordan RA, Leal S, Lo E, Tassery H, Thomson WM, Manton DJ. When to intervene in the caries process? An expert Delphi consensus statement. Clin Oral Investig. 2019 Oct;23(10):3691-3703. doi: 10.1007/s00784-019-03058-w. Epub 2019 Aug 23. PMID 31444695
- [Background] Urquhart O, Tampi MP, Pilcher L, Slayton RL, Araujo MWB, Fontana M, Guzman-Armstrong S, Nascimento MM, Novy BB, Tinanoff N, Weyant RJ, Wolff MS, Young DA, Zero DT, Brignardello-Petersen R, Banfield L, Parikh A, Joshi G, Carrasco-Labra A. Nonrestorative Treatments for Caries: Systematic Review and Network Meta-analysis. J Dent Res. 2019 Jan;98(1):14-26. doi: 10.1177/0022034518800014. Epub 2018 Oct 5. PMID 30290130
- [Background] Splieth CH, Ekstrand KR, Alkilzy M, Clarkson J, Meyer-Lueckel H, Martignon S, Paris S, Pitts NB, Ricketts DN, van Loveren C. Sealants in dentistry: outcomes of the ORCA Saturday Afternoon Symposium 2007. Caries Res. 2010;44(1):3-13. doi: 10.1159/000271591. Epub 2009 Dec 31. PMID 20068302
- [Background] Beiruti N, Frencken JE, van't Hof MA, Taifour D, van Palenstein Helderman WH. Caries-preventive effect of a one-time application of composite resin and glass ionomer sealants after 5 years. Caries Res. 2006;40(1):52-9. doi: 10.1159/000088907. PMID 16352882
- [Background] Ismail AI, Sohn W, Tellez M, Amaya A, Sen A, Hasson H, Pitts NB. The International Caries Detection and Assessment System (ICDAS): an integrated system for measuring dental caries. Community Dent Oral Epidemiol. 2007 Jun;35(3):170-8. doi: 10.1111/j.1600-0528.2007.00347.x. PMID 17518963
- [Background] Oba AA, Dulgergil T, Sonmez IS, Dogan S. Comparison of caries prevention with glass ionomer and composite resin fissure sealants. J Formos Med Assoc. 2009 Nov;108(11):844-8. doi: 10.1016/S0929-6646(09)60415-0. PMID 19933027